CLINICAL TRIAL: NCT00073229
Title: Killer Cells and Viral Load in Vertical HIV Infection
Brief Title: Immune Function of Infants With HIV
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Katherine Luzuriaga, MD, University of Massachusetts
Other Study IDs: 5R01AI032391-15 (NIH); 5R01AI032391-11 (NIH); 5R01AI032391-14 (NIH)
Record Dates: First submitted 2003-11-18; First posted 2003-11-19 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-09

CONDITIONS: HIV Infections
Keywords: AIDS; Vertical Transmission; Acute Infection
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
This observational study will evaluate data from infants born to HIV infected mothers in order to better characterize disease progression in early HIV infection.

DETAILED DESCRIPTION:
The role of HIV-specific cytotoxic T-lymphocytes (CTL) in controlling viremia and protecting against disease progression following vertical infection may be dependent upon CTL functional responses as well as on the timing of detection, magnitude, and breadth of the responses. Novel and sensitive assay systems (MHC-peptide tetramers, ELISPOT assays, intracellular cytokine assays) have enhanced the detection and characterization of virus-specific CTL responses in the peripheral blood. This study will use these novel methods to examine the timing of detection, magnitude, specificity, and in vitro functional properties of HIV-specific CTL in infants; to evaluate the effects of potent combination antiretroviral therapy on HIV-specific CTL in infants; and to evaluate the immunogenicity of recombinant pox-based vaccines in HIV infected infants with prolonged viral suppression following early potent combination antiretroviral therapy.

Blood samples from infants born to HIV infected women will be obtained from infants enrolled in other HIV trials. Generally, samples will be obtained at birth, Week 1, and Months 1, 2, 4, 6, 9, and 12.

ELIGIBILITY:
Inclusion Criteria:

* Infants and children born to HIV infected women

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2000-07; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Luzuriaga, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Background] Gibson L, Piccinini G, Lilleri D, Revello MG, Wang Z, Markel S, Diamond DJ, Luzuriaga K. Human cytomegalovirus proteins pp65 and immediate early protein 1 are common targets for CD8+ T cell responses in children with congenital or postnatal human cytomegalovirus infection. J Immunol. 2004 Feb 15;172(4):2256-64. doi: 10.4049/jimmunol.172.4.2256. PMID 14764694
- [Background] Luzuriaga K, McManus M, Mofenson L, Britto P, Graham B, Sullivan JL; PACTG 356 Investigators. A trial of three antiretroviral regimens in HIV-1-infected children. N Engl J Med. 2004 Jun 10;350(24):2471-80. doi: 10.1056/NEJMoa032706. PMID 15190139
- [Background] Obaro SK, Pugatch D, Luzuriaga K. Immunogenicity and efficacy of childhood vaccines in HIV-1-infected children. Lancet Infect Dis. 2004 Aug;4(8):510-8. doi: 10.1016/S1473-3099(04)01106-5. PMID 15288824
- [Background] Safrit JT, Ruprecht R, Ferrantelli F, Xu W, Kitabwalla M, Van Rompay K, Marthas M, Haigwood N, Mascola JR, Luzuriaga K, Jones SA, Mathieson BJ, Newell ML; Ghent IAS Working Group on HIV in Women Children. Immunoprophylaxis to prevent mother-to-child transmission of HIV-1. J Acquir Immune Defic Syndr. 2004 Feb 1;35(2):169-77. doi: 10.1097/00126334-200402010-00012. PMID 14722451
- [Background] Scott ZA, Beaumier CM, Sharkey M, Stevenson M, Luzuriaga K. HIV-1 replication increases HIV-specific CD4+ T cell frequencies but limits proliferative capacity in chronically infected children. J Immunol. 2003 Jun 1;170(11):5786-92. doi: 10.4049/jimmunol.170.11.5786. PMID 12759463
- [Result] Sanchez-Merino V, Nie S, Luzuriaga K. HIV-1-specific CD8+ T cell responses and viral evolution in women and infants. J Immunol. 2005 Nov 15;175(10):6976-86. doi: 10.4049/jimmunol.175.10.6976. PMID 16272358